CLINICAL TRIAL: NCT04130009
Title: Total Knee Arthroplasty With and Without Tourniquet: Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan4
Record Dates: First submitted 2019-10-13; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Total Knee Arthroplasty
Keywords: Thigh pain; Total knee Arthroplasty; Tourniquet

STUDY DESIGN:
Intervention Model Description: This is comparative study between two groups one treated by Total knee with tourniquet and other group without tourniquet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TKA with tourniquet (Active Comparator): This group was treated by TKA with the use of tourniquet
  Interventions: Procedure: Tourniquet use
- TKA without tourniquet (Active Comparator): This group was treated by TKA without tourniquet
  Interventions: Procedure: Tourniquet use

INTERVENTIONS:
Procedure: Tourniquet use — Use of Tourniquet in The TKA
  Other Names: No tourniquet use

SUMMARY:
Tourniquet use during total knee arthroplasty (TKA) improves visibility and reduces intraoperative blood loss. However, tourniquet use may also have a negative impact on early recovery of muscle strength and lower extremity function after TKA.Seventy Patients are involved in this study and were divided into two groups; Group A (35) patients were treated with TKA with pneumatic thigh tourniquet. Group B (35) patients were treated with TKA without tourniquet. All patients were suffering from severe knee osteoarthritis and they failed to respond to conservative treatment so they are candidates for primary TKA. The two groups are matched related to age and gender. Selection of patients into two groups done randomly with regard of odd number for group A and even number for group B

DETAILED DESCRIPTION:
This study started on March 2016 and ends on October 2018. Seventy Patients are involved in this study and were divided into two groups; Group A (35) patients were treated with TKA with pneumatic thigh tourniquet. Group B (35) patients were treated with TKA without tourniquet. All patients were suffering from severe knee osteoarthritis and they failed to respond to conservative treatment so they are candidates for primary TKA. The two groups are matched related to age and gender. Selection of patients into two groups done randomly with regard of odd number for group A and even number for group B. All patients were followed for a period of two weeks until removal of skin sutures for the following parameters:

Amount of blood transfusion done at and after surgery. Amount of blood drained postoperatively through suction drain. Occurrence of postoperative wound hematoma. VAS (Visual analogue score) for thigh pain at 1st day and (2) weeks postoperatively.

Clinical DVT.

ELIGIBILITY:
Inclusion Criteria:

* patients were suffering from severe knee osteoarthritis and they failed to respond to conservative treatment

Exclusion Criteria:

* Hb less than 12.
* D.M.,Blood dyscrasia.
* Any evidence of infection by screening test ESR and CRP. ,
* BMI more than 30.

Ages: 48 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue score for thigh pain | The VAS for thigh pain was measured in the day 14 after operation
  This is measurement of the degree of thigh pain after operation which range from zero to 10

IPD SHARING:
Plan to Share IPD: Undecided